CLINICAL TRIAL: NCT06604247
Title: The Association Between CBT-I Dose and Innate Immunity in Insomnia and Fatigue in Prostate Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 834620
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer; Prostate Cancer
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 4-session (Experimental): Participants randomized to this condition received 4 weekly CBT-I sessions.
  Interventions: Behavioral: Cognitive Behavioral therapy for insomnia (CBT-I)
- 8-session (Experimental): Participants randomized to this condition received 8 weekly CBT-I sessions.
  Interventions: Behavioral: Cognitive Behavioral therapy for insomnia (CBT-I)
- 10-session (Experimental): Participants randomized to this condition received 10 weekly CBT-I sessions.
  Interventions: Behavioral: Cognitive Behavioral therapy for insomnia (CBT-I)
- 12-session (Experimental): Participants randomized to this condition received 12 weekly CBT-I sessions.
  Interventions: Behavioral: Cognitive Behavioral therapy for insomnia (CBT-I)

INTERVENTIONS:
Behavioral: Cognitive Behavioral therapy for insomnia (CBT-I) — Cognitive Behavioral Therapy for Insomnia includes evaluation and orientation; data acquisition and delivery of sleep restriction therapy & stimulus control instructions; review of sleep hygiene; cognitive therapy [decatastrophization]; managing nonadherence and relapse prevention), and, finally, the final sessions will be largely focused on time-in-bed titration.

SUMMARY:
The objective of this project is to test the association between Cognitive Behavioral Therapy for Insomnia dose (number of sessions), severity of cancer related fatigue, and levels of innate immunity biomarkers. Ultimately, this research will help to develop a better understanding of the underlying mechanisms of cancer related fatigue.

DETAILED DESCRIPTION:
Cancer-related fatigue (CRF) and insomnia are prevalent among cancer patients and have been linked to decreases in quality of life and poorer overall survivorship. Currently, the mechanisms underlying CRF are not well understood, which has led to treatments that are only moderately effective. In addition, when compared to Cognitive Behavioral Therapy for Insomnia (CBT-I) in the general population, the treatment outcomes in CBT-I with cancer patients are subpar and, as such, this study will evaluate whether dose of CBT-I is effective in ameliorating CRF.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of organ-confined breast cancer or prostate cancer
* Received radiation treatment
* Willing and able to provide informed consent
* Endorse problem with both insomnia and cancer-related fatigue, as measured by the insomnia severity index, Multidimensional Fatigue Symptom Inventory (short form) and the Brief Fatigue Inventory

Exclusion Criteria:

* History of obstructive Sleep Apnea
* History of narcolepsy
* Night shift work
* Distant metastatic disease at presentation
* Active drug/alcohol dependence

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Fatigue | From enrollment to three months post-treatment
  Fatigue, as measured by the Multidimensional Fatigue Symptom Inventory-Short Form and the FACIT-Fatigue scale.
Insomnia Severity | From enrollment to post-treatment, and 3 months post-treatment
  As measured by the Insomnia Severity Index

SECONDARY OUTCOMES:
Sleep Continuity | From enrollment to post-treatment, and 3 months post-treatment.]
  As measured by the daily sleep diary, including sleep latency, number of awakenings, wake after sleep onset, total sleep time and sleep efficiency.

CONTACTS AND LOCATIONS:
Locations (1):
- University Of Pennsylvania, Behavioral Sleep Medicine Program, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided